CLINICAL TRIAL: NCT00910923
Title: Single Ascending Dose
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-38431055 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR015703
Record Dates: First submitted 2009-03-19; First posted 2009-06-01 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: JNJ-38431055

SUMMARY:
This will be a single center study conducted in two parts. Part 1 will assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of single ascending doses of JNJ-38431055 in healthy male volunteers. Part 2 will assess the effect of food on the pharmacokinetics of JNJ-38431055.

DETAILED DESCRIPTION:
The study includes 2 Parts and will be conducted at a single center. Part 1 is a randomized (study drug assigned by chance), double-blind (neither the volunteer or investigator knows the name of the assigned study drug), placebo-controlled (placebo is a substance that looks the same as JNJ-38431055 but contains no JNJ-38431055), single ascending dose study. In Part 1, study drug (i.e., JNJ-38431055 or placebo) will be administered orally as single doses on Day 1 or three treatment periods. In Part 1, for each volunteer, the study will consist of a screening evaluation visit, 3 periods of double-blind treatment, and a final, follow-up examination. The total study duration for each volunteer will be approximately 9 weeks. Part 2 is a randomized, open-label, 2-period crossover study to evaluate the effect of administering JNJ-38431055 together with food on the pharmacokinetics of JNJ-38431055, as compared to administration in the fasting condition. In Part 2, study drug (JNJ-38431055 will be administered orally as single doses on Day 1 or two treatment periods. There will be at least 7 days between doses. In Part 1, study drug (i.e., JNJ-38431055 or placebo) will be administered orally as single doses on Day 1 of three treatment periods. In Part 2, study drug (JNJ-38431055) will be administered orally as single doses on Day 1 of two treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.5 and 29.9 kg/m2 (inclusive)
* Healthy on the basis of physical examination including medical history, vital signs, 12-lead ECG, and all other screening lab tests performed
* Volunteers must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* History of, or currently active, illness or medical condition or disorder that the Investigator considers to be clinically significant
* Smoker or tobacco user within the past 6 months
* History of recent major surgery (within 6 months of study start)
* Positive test for alcohol and/or drugs of abuse
* Psychological and/or emotional problems, which would render the informed consent invalid, or limit the ability of the volunteer to comply with the study requirements
* Any condition that, in the opinion of the investigator, would compromise the well being of the volunteer or the study or prevent the volunteer from meeting or performing study requirements.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of JNJ-38431055

SECONDARY OUTCOMES:
To assess the pharmacodynamic effects of JNJ-38431055 on plasma glucose and insulin, during a Meal Tolerance Test (MTT)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.